CLINICAL TRIAL: NCT01744392
Title: Evaluate Changes in Medication Adherence and Patient Perspective of Polyglot Systems, Inc's Meducation Technology
Brief Title: Medication Adherence With Polyglot Meducation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 01658
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Results first posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension; Diabetes; Hypercholesterolemia
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Hypercholesterolemia | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- education intervention (Experimental): The intervention provides a personalized Meducation calendar to all patients enrolled in the study (identified in package as Example Calendar). The Meducation Calendar will include medications for diabetes (sugar), high blood pressure, cholesterol, heart medications and blood thinning medications. The medication calendars contains the following for each medication 1) the name, 2) the time of day, including a pictorial display, it should be taken 3) the number of times each day to take the medication, and 4) the indication for the medication.
  Interventions: Behavioral: education intervention

INTERVENTIONS:
Behavioral: education intervention — Each patient will receive instructions on how to use the medication calendar to help them adhere to their medication regimen. The Meducation Calendar is developed by the clinical pharmacist participating in the research study). The clinical pharmacist will enter the medication regimen for each participant into the application for Meducation Calendar Development.

SUMMARY:
The investigators propose a 6 month pre-post, pilot,feasibility study with up to 25 individuals among veterans with cardiovascular disease risk factors including Hypertension (HT), Diabetes Mellitis (DM) and Hyperlipidemia (HL) who receive care from the hospital-based primary care clinics associated with Durham VAMC. The investigators will examine veteran's perception and ease of using an innovative tool to help improve medication adherence to cardiovascular medications. This study aims to focus on patients with multiple chronic conditions and their caregivers to address 1) appropriate use of medications 2)maximize patient self-care and care by families and other caregivers 3) make available a tool for medication management 4) managing complex regimens, and 5) addressing health literacy.

DETAILED DESCRIPTION:
Recruitment letter:

Each week, the research assistant (RA) will identify participants who have a medical appointment scheduled 3 weeks from the current date from the statistician's list of eligible participants. The RA will review Computerized Patient Record System (CPRS) to confirm enrollment at the Durham VA Medical Center (DVAMC) or Raleigh Community Based Outpatient Clinic (CBOC), identify participants' primary care provider and conduct a preliminary medical record review of the exclusion criteria listed above.

An introductory recruitment letter signed by the patient's provider will be sent to these participants.

Telephone Screening:

The RA will call the participants between 1 and 2 weeks later to assess interest and eligibility using the telephone screening script. During this telephone call, the RA will ask permission to conduct the telephone screening to further evaluate the participants' eligibility to participate in the study. These screening questions are being asked because exclusion criteria may not be accurately reflected in the VA medical record. If participants agree to meet with study team to further discuss the project they will be scheduled for an interview. If requested, participant will be sent an appointment reminder letter signed by the study principal investigator and/or project coordinator.

All participants will be sent reminder letters up to 3 weeks prior to their scheduled 3 and 6 month follow-up appointments.

Consent Process:

At this interview, the patient will be given greater detail about the study, and if agreeable, will provide written informed consent. Participants who consent to participate in the study and agree to be digitally audio recorded will also have complete form 10-3203 "Consent for use of picture and /or voice" at baseline.

Interview Procedures:

RAs will obtain the participants' outcome values (i.e., BP) from the clinical record at baseline, at 3 month follow-up. This information will be double-entered into an application on the Health Services Research & Development (HSRD) VA Server. At baseline and 3-month follow-up contacts, participants will also undergo an interview to determine secondary outcome variables including self-reported medication adherence and perceptions of the intervention. The baseline interview will be conducted in person if possible, however, at the 3 month follow-up appointment the interview will be conducted by telephone. The RA's will work with patients to be seen in a 6 week window around the original follow-up appointment. Pill refill will be calculated for all individuals at 6 months.

Participant Contacts In-person meeting - Baseline After the consent process, at the baseline interview, a research assistant(RA) will conduct the outcome assessment procedures, which includes asking the participant questions about their age,race, medical history, self reported adherence to cardiovascular medications and their understanding about the risk of cardiovascular disease. The RA will also ask questions about their lifestyle, and quality of life. Participants who qualify for enrollment and provide informed consent will meet with the research pharmacist for education use of the Meducation Calendar.

3 month follow-up interview. A research assistant will contact participant via phone to determine secondary outcome variables including self reported medication adherence to cardiovascular medications. The entire interview should take no more than 30 minutes.

Optional Qualitative: 3 month phone interview: For selected intervention participants only the RA will conduct a questionnaire about the participant's perception to determine which aspects of the Meducation Calendar intervention were most helpful for participants and which aspects need revision. Participants who agreed to the qualitative interview during the consent process will be asked during the 3 month interview to confirm their continued desire to participate in the audio recorded phone interview if selected. This visit should take no more than 30 minutes. Those selected to participate will be scheduled to complete the qualitative interview over the phone within 15 days from the time they complete the intervention and interview. The qualitative interview will be audio recorded digitally on a VA owned and configured computer and later transcribed using VA owned computer software. Names will not be associated with the audio recordings. After all recordings have been analyzed and coded, recordings will be destroyed in accordance with VA Information Security procedures. This phone call for the optional qualitative interview should take no more than 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in one of three DVAMC Primary Care Clinics affiliated with the hospital for at least one year;
* At least one visit to a primary care provider (PCP) at Durham VAMC associated primary care clinics in the previous 12 months;
* Outpatient diagnostic code for hypertension (> 140/90), diabetes and/or hypercholesterolemia
* Prescription for metoprolol tartrate (twice a day beta blocker, most common 2 day medication prescribed in the VA)
* Baseline Medication Possession Ratio (MPR) of < 80% indicating medication non adherence
* More than 9 active medications.

Exclusion Criteria:

* diagnosed with metastatic cancer,
* diagnosed with dementia documented in medical record,
* active diagnosis of psychosis documented in medical record with admission with last 30 days
* participating in another clinical trial,
* not currently receiving care at the Durham VAMC
* resident of a nursing home,
* hard time seeing type/printing on books, magazines articles, etc.
* hard time hearing or speaking on the telephone
* limited/no access to telephone
* currently a patient in the primary care pharmacist medication management clinic at Durham VAMC
* plans to move medical care from DVAMC in next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hayden B Bosworth, PhD, Principal Investigator — Durham VA Medical Center
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Education Intervention
Started | 23
Completed | 22
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Education Intervention
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 21
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 9
  African American | 14
Region of Enrollment [Number; unit: participants]
  United States | 23
Health Literacy [Number; unit: participants] — Health Literacy is measured using the Rapid Assessment of Adult Literacy in Medication, a 66-item word recognition evaluation.The REALM scores range from 0 - 66, with scores from 0-18 consistent with <= 3rd grade health literacy, 19-44 = 4th - 6th grade, 45-60 = 7th - 8th grade, 61-66 >= 9th grade. For the purposes of this study Low Health Literacy is defined as a REALM score <60 vs High Health Literacy as a REALM score >= 61.
  participants
    Low Health Literacy | 9
    High Health Literacy | 14
Employed (full or part-time) [Number; unit: participants]
  Employed | 7
  Not Employed | 16

OUTCOME MEASURES:

1. Primary Outcome: Medication Possession Ratio at Baseline
Description: Medication Possession Ratio (MPR) is defined as the number of daily doses of medication dispensed by the pharmacy to each patient, divided by the patient's total follow-up time." The time period for the assessment for baseline MPR 12 months prior to enrollment.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percentage of medication possession
Groups:
- Education Intervention: The intervention provides a personalized Meducation calendar to all patients enrolled in the study. The Meducation Calendar includes medications for diabetes (sugar), high blood pressure, cholesterol, heart medications and blood thinning medications. The medication calendars contains the following for each medication 1) the name, 2) the time of day, including a pictorial display, it should be taken 3) the number of times each day to take the medication, and 4) the indication for the medication. Each patient will receive instructions on how to use the medication calendar to help them adhere to their medication regimen. The Meducation Calendar is developed by the clinical pharmacist participating in the research study. The clinical pharmacist will enter the medication regimen for each participant into the application for Meducation Calendar Development.
Arm/Group | Education Intervention
Number analyzed (Participants) | 23
percentage of medication possession | 65.0 (1.14)

2. Primary Outcome: Medication Possession Ratio at 6 Months
Description: Medication Possession Ratio (MPR) is defined as the number of daily doses of medication dispensed by the pharmacy to each patient, divided by the patient's total follow-up time." The time period for the assessment for 6 months MPR 6 months after enrollment.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of medication possession
Arm/Group | Education Intervention
Number analyzed (Participants) | 23
percentage of medication possession | 68.2 (0.28)
Statistical Analysis 1: Comparison: Education Intervention; Difference between percentages. Increases in value indicate improvement in adherence; Test type: Superiority or Other; p = .73, t-test, 2 sided; Mean Difference (Final Values) = 3.2

3. Secondary Outcome: Blood Pressure at Baseline
Description: Clinical Characteristics at Baseline for Systolic & Diastolic Blood Pressure,
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Education Intervention
Number analyzed (Participants) | 23
mmHg
  Systolic Blood Pressure | 130.06 (15.1)
  Diastolic Blood Pressure | 76.6 (8.0)

4. Secondary Outcome: Blood Pressure at 6 Months
Description: Clinical Characteristics at 6 months for Systolic & Diastolic Blood Pressure,
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Education Intervention
Number analyzed (Participants) | 23
mmHg
  Systolic Blood Pressure | 130.1 (18.4)
  Diastolic Blood Pressure | 75.1 (10.4)

5. Secondary Outcome: Cholesterol & Creatinine Levels at Baseline
Description: Clinical Characteristics at Baseline for LDL, HDL,Total Cholesterol and Creatinine
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Education Intervention
Number analyzed (Participants) | 23
mg/dL
  LDL Cholesterol | 77.0 (17.4)
  HDL Cholesterol | 45.1 (19.5)
  Total Cholesterol | 152.4 (41.4)
  Creatinine | 1.1 (0.2)

6. Secondary Outcome: Cholesterol & Creatinine Levels at 6 Months
Description: Clinical Characteristics at 6 months for LDL, HDL,Total Cholesterol and Creatinine
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Education Intervention
Number analyzed (Participants) | 23
mg/dL
  LDL Cholesterol | 82.3 (16.9)
  HDL Cholesterol | 46.4 (26.1)
  Total Cholesterol | 160.0 (41.7)
  Creatinine | 1.2 (0.3)

7. Secondary Outcome: Weight at Baseline
Description: Clinical Characteristics at Baseline for Weight
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Education Intervention
Number analyzed (Participants) | 23
pounds | 223.0 (2.9)

8. Secondary Outcome: Weight at 6 Months
Description: Clinical Characteristics at 6 months for Weight
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Education Intervention
Number analyzed (Participants) | 23
pounds | 219.4 (48.9)

9. Secondary Outcome: Pulse at Baseline
Description: Clinical Characteristics at Baseline for Pulse
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Education Intervention
Number analyzed (Participants) | 23
beats per minute | 73.2 (20.9)

10. Secondary Outcome: Pulse at 6 Months
Description: Clinical Characteristics at 6 month for Pulse
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Education Intervention
Number analyzed (Participants) | 23
beats per minute | 70.3 (14.0)

ADVERSE EVENTS:
Time Frame: From enrollment through study completion (6 months)
Arm/Group | Education Intervention
Serious Adverse Events (participants affected / at risk) | 14/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Education Intervention (N=23)
Infections (Infections and infestations) | 3 (3)
ER visit (Injury, poisoning and procedural complications) | 1 (1)
Vascular Event (Vascular disorders) | 2 (2)
ER visit (Psychiatric disorders) | 1 (2)
ER visit (Respiratory, thoracic and mediastinal disorders) | 2 (3)
ER visit (General disorders) | 3 (3)
Hospitalization (Cardiac disorders) | 2 (2)
ER visit (Musculoskeletal and connective tissue disorders) | 3 (3)
ER (Gastrointestinal disorders) | 2 (2)
Hospitalization (Renal and urinary disorders) | 1 (1)
ER Visit (Endocrine disorders) | 1 (1)
Hospitalization (Nervous system disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No